CLINICAL TRIAL: NCT02649647
Title: Randomized Trial of Sphincter-Preserving Surgery With Proximally Extended Resection Margin on Bowel Function and Anastomotic Complication for Rectal Cancer Patients After Neoadjuvant Chemoradiotherapy
Brief Title: Proximally Extended Resection for Rectal Cancer After Neoadjuvant Chemoradiotherapy
Acronym: PERN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Shanghai Changzheng Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERN2015019
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Neoadjuvant therapy; Chemoradiotherapy; Resection margin; Bowel function; Anastomosis
MeSH Terms: conditions — Rectal Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Resection (Active Comparator): Patients receive conventional resection with standard proximal excision margin. The sigmoid colon is anastomosed to the rectum or anus. A defunctioning ileostomy is routinely performed.
  Interventions: Procedure: Conventional resection
- Proximally Extended Resection (Experimental): Patients receive proximally extended resection. The whole sigmoid colon and rectum proximal to the tumor is removed, and the descending colon is anastomosed to the rectum or anus. A defunctioning ileostomy is routinely performed.
  Interventions: Procedure: Proximally extended resection

INTERVENTIONS:
Procedure: Conventional resection — The conventional technique requests an excision of at least 10 cm of bowel proximal to the tumor, and the sigmoid colon is anastomosed to the rectum or anus. A defunctioning ileostomy is routinely performed.
  Arms: Conventional Resection
Procedure: Proximally extended resection — The modified technique requests an excision of the whole sigmoid colon and rectum proximal to the tumor, and the descending colon is anastomosed to the rectum or anus. A defunctioning ileostomy is routinely performed.
  Arms: Proximally Extended Resection

SUMMARY:
Neoadjuvant chemoradiotherapy has been recommended as the standard preoperative treatment for locally advanced rectal cancer. However, preoperative radiotherapy increases the risk of bowel dysfunction after sphincter-preserving surgery, for which patients suffer from incontinence, urgency, and unpredictability defecation problems. Furthermore, preoperative chemoradiotherapy is a potential risk factor of anastomotic leakage and stenosis after rectal cancer surgery.

Unhealthy anastomosis, with both ends of injured bowel segments after pelvic radiation, is a major concern. When conventional surgical procedures would retain part of sigmoid colon that has been included in the radiation target, sphincter-preserving surgery with proximally extended resection margin could provide an intact proximal colon limb for the anastomosis.

It is not known yet whether proximally extended resection improves postoperative bowel function or anastomotic integrity for patients with rectal cancer after neoadjuvant chemoradiotherapy. The proposed study will compare sphincter-preserving surgery with and without proximally extended resection margin, to observe the postoperative bowel function, as well as the incidence of anastomotic complication. This study will examine a new surgical strategy, which potentially benefits the patients undergoing neoadjuvant chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* ECOG performance status: 0-2
* Histologically confirmed adenocarcinoma of the rectum
* Distal border of the tumor located ≤ 12 cm from the anal verge
* Primary stage T3-4 or any node-positive disease
* Undergoing long-course 5-fluorouracil based neoadjuvant chemoradiotherapy
* Conventional fractionated radiotherapy of at least 45 Gy
* Resectable disease after neoadjuvant chemoradiotherapy
* No evidence of distant metastasis
* Amenable to sphincter-preserving surgery
* Tolerable to general anesthesia
* Provision of written informed consent

Exclusion Criteria:

* Prior or concurrent malignancies within the past 5 years except for effectively treated squamous cell or basal cell skin cancer, melanoma in situ, or carcinoma in situ of the cervix
* Synchronous colon cancer
* History of colorectal resection except appendectomy
* Acute intestinal obstruction or perforation
* Multiple visceral resection
* Abdominoperineal resection
* American Society of Anesthesiologists (ASA) class Ⅳ or Ⅴ
* Pregnant or nursing, fertile patients do not use effective contraception
* Serious cardiovascular disease, uncontrolled infections, or other serious uncontrolled concomitant disease
* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-02; Primary Completion 2024-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of major bowel dysfunction | at the time of 12 months after the restoration of defunctioning stoma
  Low anterior resection syndrome score (LARS score) will be used to assess the bowel function. Number of participants with major LARS will be calculated for the incidence of major bowel dysfunction.

SECONDARY OUTCOMES:
Incidence of anastomotic leakage | up to 6 months postoperatively
Incidence of anastomotic stenosis | 12 months postoperatively
Incidence of major bowel dysfunction | at the time of 36 months after the restoration of defunctioning stoma
  Low anterior resection syndrome score (LARS score) will be used to assess the bowel function.
Incidence of major bowel dysfunction | at the time of 60 months after the restoration of defunctioning stoma
  Low anterior resection syndrome score (LARS score) will be used to assess the bowel function.
3-year disease free survival | 3 years
5-year overall survival | 5 years
Incidence of anastomotic haemorrhage | up to 1 month postoperatively
Incidence of intraoperative complication | at the time of surgery
Postoperative morbidity | up to 30 days postoperatively
Postoperative mortality | up to 30 days postoperatively
Quality of life impairment | at the time of 12 months after the restoration of defunctioning stoma
  Quality of life will be assessed by EORTC QLQ-C30 and EORTC QLQ-CR29.
Quality of life impairment | at the time of 36 months after the restoration of defunctioning stoma
  Quality of life will be assessed by EORTC QLQ-C30 and EORTC QLQ-CR29.
Quality of life impairment | at the time of 60 months after the restoration of defunctioning stoma
  Quality of life will be assessed by EORTC QLQ-C30 and EORTC QLQ-CR29.

OTHER OUTCOMES:
Incidence of major bowel dysfunction in patients with tumor of different location | at the time of 12 months after the restoration of defunctioning stoma
Incidence of major bowel dysfunction in patients with tumor of different location | at the time of 36 months after the restoration of defunctioning stoma
Incidence of major bowel dysfunction in patients with tumor of different location | at the time of 60 months after the restoration of defunctioning stoma
Incidence of anastomotic complication in patients with tumor of different location | up to 12 months postoperatively
Operative duration by minutes | at the time of surgery
Intraoperative blood loss by millilitres | at the time of surgery
Postoperative rehabilitation time | up to 1 months postoperatively
Postoperative hospital stay by days | up to 1 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, MD, PhD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University; Hui Wang, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China